CLINICAL TRIAL: NCT01452087
Title: Health Benefits of Chronic vs. Acute Exercise in Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, JEFFREY F HOROWITZ, Associate Professor, Movement Science, School of Kinesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01 DK077966 - R; R01DK077966 (NIH)
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Obesity
Keywords: insulin sensitivity; exercise
MeSH Terms: conditions — Obesity; Insulin Resistance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise Session (Other): Subjects will exercise on a treadmill for 1 hour at moderate intensity (i.e., 90% of the exercise intensity found to elicit their ventilatory threshold during the preliminary testing, which is equivalent to approximately 60% of their maximal predicted heart rate).
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Subjects will exercise on a treadmill for 1 hour at moderate intensity (i.e., 90% of the exercise intensity found to elicit their ventilatory threshold during the preliminary testing, which is equivalent to approximately 60% of their maximal predicted heart rate).

SUMMARY:
Compare the effects of single session of exercise vs. chronic exercise training on key risk factors associated with Metabolic Syndrome (e.g., glucose tolerance, blood lipid profile, and blood pressure) in overweight adults.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 27-34 kg/m2;
* Regular exercisers(≥4 days/wk of aerobic exercise;
* 30-60min/session at moderate and vigorous intensities);
* Non-exercisers (no regularly planned exercise/physical activity);
* Women must have regularly occurring menses and must be premenopausal.

Exclusion Criteria:

* Pregnant or lactating;
* Evidence/history of cardiovascular or metabolic disease;
* Currently taking medications known to affect lipid or glucose metabolism.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2009-05; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
oral glucose tolerance test | 2 hour

SECONDARY OUTCOMES:
Resting Metabolic Rate | 20-30 min

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Substrate Metabolism Laboratory, Ann Arbor, Michigan, United States